CLINICAL TRIAL: NCT05950386
Title: Effects of Lead Exposure on Iron Metabolism and the Nrf2-dependent Ferroptosis Pathway
Brief Title: Effects of Lead Exposure on Ferroptosis Pathway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northern Jiangsu People's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, WenJing Zhao, Principal Investigator, Northern Jiangsu People's Hospital
Other Study IDs: Lead exposure
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lead Poisoning; Neurotoxicity
Keywords: Ferroptosis; Nrf2; Iron metabolism; Lead exposure; Neurotoxicity
MeSH Terms: conditions — Lead Poisoning; Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The enrolled participant's peripheral whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The control group: The invited non-lead-exposed workers live in Yangzhou, Jiangsu, China
- The lead exposure group: The invited chronic-lead exposed workers live in Yangzhou, Jiangsu, China
  Interventions: Other: Lead exposure

INTERVENTIONS:
Other: Lead exposure — The lead-acid battery factory workers will exposure to lead via Inhalation of lead particles, ingestion of lead-contaminated dust and water.
  Groups: The lead exposure group

SUMMARY:
The aim of this study was to investigate the effects of chronic lead exposure on iron metabolism and the Nrf2-dependent ferroptosis pathway in lead acid battery factory workers

DETAILED DESCRIPTION:
Background:

Lead (Pb) is a prevalent and highly toxic heavy metal. Human activities have been the primary cause of lead contamination in the environment over the past century. Lead exposure poses a global concern, particularly for children, and individuals can be exposed to lead through various means, such as contaminated soil, dust, food, water, or foreign objects. The central nervous system (CNS) is particularly vulnerable to the toxic effects of lead (Pb), especially in children, primarily due to the immaturity of the blood-brain barrier.

Ferroptosis is a recently defined form of regulated cell death characterized by iron-dependent cell death resulting from the accumulation of lipid hydroperoxides. However, the exact mechanism underlying the neurotoxic effects of chronic low-level lead exposure-induced ferroptosis on neuronal injury is not yet fully understood.

Methods:

The investigators first analyze the difference of blood lead level using atomic absorption spectrometry.

The investigators enrolled 20 chronic lead exposure workers from a lead acid battery factory and an age-matched control group of non-lead-exposed workers.

TNF-α elisa kit was used to compare the proinflammatory cytokines in two groups.

Quantitative reverse transcription PCR (Polymerase Chain Reaction) was used to compare messenger ribonucleic acid (mRNA) expression of iron metabolism (FTH1, FPN1, DMT1) and the Nrf2-dependent ferroptosis pathway (Nrf2, SLC7A11, GPX4)

Detailed Methods protocol

1. The criteria of enrolled chronic lead exposure participants were as follows：inclusion: work for this lead acid battery factory more than 10 year; exclusion: exposure to any chemistry pollution before; neurological disorders; endocrine diseases; cancer
2. Sample collection: at the end of recruitment in this study, all of the enrolled participant will come to the hospital to collect peripheral Blood (Northern Jiangsu People's Hospital, affiliated with Yangzhou University), and the blood samples will be collected into EDTA (ethyleneDiamine tetraacetic acid) vacutainer tubes and then divided into leukocytes and plasma for further experiments.
3. TNF-α ELISA KIT: Plasma TNF-α concentrations were detected by the competitive ELISA method
4. Primer sequence used in this study:

1.DMT1 forward: 5'-CTAGACTGGGAGTGGTTACTGG-3' DMT1 reverse: 5'-AGGATGACTCGTGGGACCTT-3' 2.FTH1 forward: 5'-CTGGTGGCCGAATCTTCCTTCA-3' FTH1 reverse: 5'-GCCAGTTTGTGCAGTTCCAG-3' 3.FPN1 forward: 5'-CTACTTGGGGAGATCGGATGT-3' FPN1 reverse: 5'-CTGGGCCACTTTAAGTCTAGC-3' 4.GPX4 forward: 5'-GAGGCAAGACCGAAGTAAACTAC-3' GPX4 reverse: 5'-CCGAACTGGTTACACGGGAA-3' 5.SLC7A11 forward: 5'-TCTCCAAAGGAGGTTACCTGC-3' SLC7A11 reverse: 5'-AGACTCCCCTCAGTAAAGTGAC-3' 6. Nrf2 forward 5'-ATAGCTGAGCCCAGTATC-3' Nrf2 reverse 5'- CATGCACGTGAGTGCTCT-3' 7. GAPDH forward: 5'-GGAGCGAGATCCCTCCAAAAT-3' GAPDH reverse: 5'-GGCTGTTGTCATACTTCTCATGG-3'

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years old
2. Work for the lead acid battery factory more than 10 years

Exclusion Criteria:

1. Neurological disorders
2. Endocrine diseases
3. Cancer
4. Exposure to any chemical pollutant before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will be selected from the invited who live in Yangzhou city via the website, email, and poster.
  The lead exposure group will be selected from the invited volunteers who live in Yangzhou with the assistance of the Center for Disease Control and Prevention of Yangzhou, the website, email, and poster.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Concentration of TNF-α level in peripheral blood | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 60 days
  Biomarkers of the proinflammatory cytokines
The relative mRNA expression rate of the Nrf2- dependent ferroptosis genes in peripheral blood | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 60 days
  Biomarkers of the Nrf2- dependent ferroptosis
The relative mRNA expression rate of the iron metabolism genes in peripheral blood | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 60 days
  Biomarkers of the iron metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Wenjing Zhao, Yangzhou, Jiangsu, China